CLINICAL TRIAL: NCT00848887
Title: A Phase Ib, Randomized, Observer-Blind, Multicenter, Factorial-Design Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Injections of Trivalent Inactivated Influenza Vaccine With or Without a Second Influenza B Strain in Combination With or Without One of Three Different Doses of Adjuvant in Healthy Children, Aged 6 to <36 Months
Brief Title: A Dose Ranging Study Comparing Different Combinations of Adjuvanted and Non-adjuvanted Influenza Vaccines in Healthy Children 6 to <36 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: V104P2; 2008-002602-20
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Influenza
Keywords: Influenza; Flu; Vaccine; Adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Adjuvanted and un-adjuvanted influenza vaccines

INTERVENTIONS:
Biological: Adjuvanted and un-adjuvanted influenza vaccines — 16 different formulations of trivalent influenza vaccine and 1 marketed influenza vaccine comparator.

SUMMARY:
This study will evaluate the safety and immunogenicity of different combinations of influenza vaccine in healthy young children.

ELIGIBILITY:
Inclusion Criteria:

* Children of 6 month to <36 month of age in good health as determined by medical history, physical assessment and clinical judgement of the investigator.

Exclusion Criteria:

* History of serious disease. History of serious reaction following administration of vaccine or hypersensitivity to vaccine components. Known or suspected impairment/alteration of immune function.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Assessment of all adverse events from time of vaccination through study end will be collected to for safety assessment. | 50 days

SECONDARY OUTCOMES:
Strain-specific influenza antibody titers will be used to assess Immunogenicity | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- UCL St. Luc - Pharmacy, Brussels, Belgium

REFERENCES:
- [Result] Della Cioppa G, Vesikari T, Sokal E, Lindert K, Nicolay U. Trivalent and quadrivalent MF59((R))-adjuvanted influenza vaccine in young children: a dose- and schedule-finding study. Vaccine. 2011 Nov 3;29(47):8696-704. doi: 10.1016/j.vaccine.2011.08.111. Epub 2011 Sep 9. PMID 21906647